CLINICAL TRIAL: NCT03370601
Title: Evaluation of the Clinical and Immunological Impact of Two Therapeutic Strategies (Increasing the Infliximab Dose or Introduction of Immunosuppressive Therapy) in Patients Chronic Inflammatory Bowel Diseases in Loss of Response to Infliximab
Brief Title: Evaluation of the Clinical and Immunological Impact of Two Therapeutic Strategies in Chronic Inflammatory Diseases
Acronym: STAMP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough recruitment Lack of funding CR
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015_23; 2015-A00940-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: crohn's disease; ulcerative colitis; infliximab; loss of response
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab; Mercaptopurine; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimisation strategy (Other): increase of Infliximab dose from 5mg/kg every 8 weeks to Infliximab 10 mg/kg every 8 weeks
  Interventions: Drug: Infliximab
- Addition strategy (Other): same dose of Infliximab ( 5mg/kg every 8 weeks) with addition of immunosuppressive agent: Azathioprine or Mercaptopurine
  Interventions: Drug: Mercaptopurine; Drug: Azathioprine; Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab 10mg/kg every 8 weeks
  Arms: Optimisation strategy
Drug: Mercaptopurine — 6-mercaptopurine 1 à 1,5 mg/kg
  Other Names: addition strategy with 6-mercaptopurine in second intention
  Arms: Addition strategy
Drug: Azathioprine — Azathioprine 2 à 2.5mg/kg/j
  Other Names: addition strategy with azathioprine in first intention
  Arms: Addition strategy
Drug: Infliximab — Infliximab 5mg/kg every 8 weeks
  Arms: Addition strategy

SUMMARY:
This study evaluates 2 therapeutic strategies (increase infliximab dose or add an immunosuppressant) in patients with inflammatory bowel disease in loss of response to infliximab. Addition of an immunosuppressant may be more efficient at long term and is less expensive.

ELIGIBILITY:
Inclusion Criteria:

* patients with ulcerative colitis or crohn's disease
* treated with infliximab (5mg/kg per 8 weeks) and with loss of response after at least 4 infusions of infliximab
* active disease ( HBI > 5 for CD patients or SCCAI> 6 for UC patients)
* patients treated with infliximab only at the time of loss of response

Exclusion Criteria:

* Patients with CD with ano perineal lesions and without luminal activity
* patients treated with cortico steroids and having had history of intolerance to azathioprin, 6-mercaptopurine or methotrexate
* patients with acute severe flare (HBI>12 for CD patients and Lichtiger score > 10 for UC patients)
* pregnant female
* patients with anal disease alone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of patients in Clinical remission | At Week 52
  the clinical remission is defined by Harvey Bradshaw (HBI) Index < 4 for Crohn's disease or Simple Clinical Colitis Activity Index (SCCAI)<4 for ulcerative colitis.

SECONDARY OUTCOMES:
Number of patients in deep remission | At Week 52
  clinical remission associated with endoscopic remission (CDEIS <3 for CD patients or Mayo score<2 for UC patients)
Number of patient in remission and clinical response | At week 16
  clinical response is defined as a decrease of at least 3 points of HBI for CD patients or SCCAI for UC patients compared to baseline (week 0).
  Simple Clinical Colitis Activity Index (SCCAI)<4 for ulcerative colitisHBI pour MC et SCCAI pour RCH <4 associated at CRP < 5 mg/dl.
infliximab blood concentration | Baseline, week 16 ad week 52
infliximab antibodies concentration | Baseline, week 16 ad week 52
economic criteria | At week 52
  medical fees in each arm
number of patient with adverse effects and allergic reactions with infliximab | At week 52
Inflammatory bowel disease questionnaire (score IBDQ) | Baseline and week 52
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Pariente, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523